CLINICAL TRIAL: NCT05254847
Title: Capecitabine Combined With Lenvatinib and Tislelizumab as Adjuvant Treatment After Resection in Patients With Biliary Tract Cancer: A Single-arm, Phase II Study
Brief Title: Capecitabine Combined With Lenvatinib and Tislelizumab as Adjuvant Treatment After Resection in Patients With BTC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Head of liver surgery department, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTC-CaLenT
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — lenvatinib; tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combined treatment group (Experimental): Capecitabine combined with lenvatinib and tislelizumab: Lenvatinib,8mg po. qd.Tislelizumab,200mg iv. q3w. Capecitabine 1250mg/m^2 bid.d1-d14 q3w
  Interventions: Drug: Capecitabine combined with lenvatinib and tislelizumab

INTERVENTIONS:
Drug: Capecitabine combined with lenvatinib and tislelizumab — Capecitabine combined with lenvatinib and tislelizumab

SUMMARY:
This is a prospective, open-label, single-center clinical study, to evaluate the efficacy and safety of Capecitabine combined with Lenvatinib and Tislelizumab as adjuvant treatment after resection in patients with biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 and above
2. Pathological reported showed Biliary tract cancer (include intrahepatic cholangiocarcinoma (IHCC), extrahepatic/hilar cholangiocarcinoma, muscle infiltrated gallbladder carcinoma or distal cholangiocarcinoma)，patients received R0 resection(including liver resection, pancreatectomy, or both).
3. ECOG PS 0-1
4. Patients can tolerate the combination therapy and survive longer than 6 months.
5. Organ function(Exclude use blood components and cell growth factors for 14 days): Neutrophils (ANC) ≥1,500/mm3, Platelet count (PLT)≥100,000/mm3, Hemoglobin (Hb) ≥9g/dL; Serum creatinine(SCR) ≤1.5*upper limit of normal(ULN),or creatinine clearance rate≥50 ml/min(Cockcroft-Gault Formula),Total bilirubin(TBIL)≤ 2*ULN,Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 3*ULN, urine protein≤2+(if urine protein≥2+, 24-hour urinary protein quantity must ≤1g), Adequate surgical biliary drainage and no infection signal.
6. The coagulation function was normal (without active bleeding and thrombotic disease): International normalized ratio(INR)≤1.5*ULN, activated partial thromboplastin time(APTT)≤1.5×ULN, prothrombin time(PT)≤1.5*ULN.
7. Women without surgical sterilization or childbearing age who are required to use a medically approved contraceptive method (such as an intrauterine device, birth control pill or condom) during the study period and for 3 months after the study period; Women are of reproductive age and not undergoing surgical sterilization whose the serum or urine HCG test must be negative within 7 days prior to study enrollment and must be non lactation period. Male patients without surgical sterilization or reproductive age are required to consent with their spouse to use a medically approved contraceptive method during the study treatment period and for 3 months after the study treatment period.
8. The patients are voluntarily enrolled in the study, with good compliance and coordinate the follow-up for safety and survival

Exclusion Criteria:

1. Patients with pancreatic/ampullary carcinoma
2. Patients with mucous gallbladder carcinoma
3. Patients who had received radiotherapy or chemotherapy previously
4. Incomplete surgery recovery or biliary obstruction exist
5. Patients with radiographs confirmed distant metastases
6. Patients with prior or concurrent malignancy(excluded Cured basal cell carcinoma of the skin and Carcinoma in situ elsewhere)
7. Patients are allergy to macromolecular protein preparation(including anti-PD-1 antibody, uracil, cytosine pharmaceutical ingredients)
8. There are significant factors affecting oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction
9. Patients had any active autoimmune disease or had experience of autoimmune disease.
10. Patients are receiving immunosuppressant and continue using within 2 weeks before enrollment
11. Patients with ascites or pleural effusion requiring therapeutic puncture or drainage
12. Patients with disease of the heart that are not well controlled
13. Abnormal coagulation(have tendency to bleed or receiving thrombolytic or anticoagulant therapy)
14. Patients had active infection or unexplained fever during screening and before first dose
15. Patients had abdominal fistula, gastrointestinal perforation, or abdominal abscess less than 4 weeks before first dose.
16. Patients past or present with pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severely impaired lung function, etc
17. Patients have congenital or acquired immune deficiency; Hepatitis B patients: HBV DNA≥10^3/ml, Hepatitis C patients: HCV RNA≥10^3/ml, Chronic hepatitis B virus carriers: HBV DNA<2000 IU/ml（<10^4 copies/ml), patients must receive antiviral therapy during the trial
18. Patients are participating in other relevant clinical studies or it has been less than 1 month since the end of the previous clinical study; Patients maybe receive other systemic antitumor therapy during the study period;
19. Patients received live vaccination less than 4 weeks before administration or possibly receive during the study period.
20. Patients had history of psychotropic substance abuse, alcohol abuse, or drug abuse.
21. Patients cannot or does not agree to pay the cost of examination and treatment expense
22. The researchers concluded the patients should be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
1 year DFS rate | 12 month
  one year disease free survival rate

SECONDARY OUTCOMES:
2 years DFS rate | 24 month
  two years disease free survival rate
1 year OS rate | 12 month
  one year overall survival rate
3 years OS rate | 36 month
  three years overall survival rate
AE | 30 days from the beginning of treatment to the last treatment
  adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

REFERENCES:
- [Derived] Feng Y, Zhang N, Zhao YM, Pan Q, Mao AR, Zhu WP, Zhang T, Wang L. Adjuvant tislelizumab, lenvatinib, and capecitabine for resected biliary tract cancer: a prospective phase II trial. BMC Med. 2026 Jan 23. doi: 10.1186/s12916-026-04650-0. Online ahead of print. PMID 41578300